CLINICAL TRIAL: NCT00163046
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, 28-day, Polysomnographic Study of Gabapentin 250 mg in Transient Insomnia Induced by a Sleep Phase Advance
Brief Title: A 28-Day Polysomnographic Study of Gabapentin in Transient Insomnia Induced by a Sleep Phase Advance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A9451155
Record Dates: First submitted 2005-09-08; First posted 2005-09-13 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2008-04

CONDITIONS: Transient Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gabapentin (Experimental)
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 250 mg oral capsule 30 minutes prior to bedtime for 28 days
  Arms: Gabapentin
Drug: Placebo — Matched placebo 30 minutes prior to bedtime for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to to assess the effect of gabapentin compared to placebo on sleep, using polysomnography along with subjective sleep assessments, in subjects with transient insomnia induced by a sleep phase advance.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older with occasional sleeplessness in the month prior to screening

Exclusion Criteria:

* Current treatment for, or recent history (within 2 years) of, a sleeping disorder including excessive snoring, obstructive sleep apnea or a chronic painful condition that interferes with the subject's sleep
* Currently taking or expected to take any of the following during trial: amphetamines, benzodiazepines, cocaine, marijuana, methaqualone, methadone, opiates, propoxyphene, barbiturates, and phencyclidine during their participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2005-10; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Polysomnographic (PSG) measurement of Wake after Persistent Sleep Onset (WAPSO) | Day 1

SECONDARY OUTCOMES:
PSG WAPSO | Day 28
PSG Latency to Persistent Sleep (LPS) | Days 1 and 28
PSG Sleep Onset Latency (SOL) | Days 1 and 28
PSG Number of Awakenings (NAW) | Days 1 and 28
PSG Wake after Sleep Onset (WASO) | Days 1 and 28
PSG Total Wake Time (TWT) plus Stage 1 Sleep | Days 1 and 28
PSG Wake Time During Sleep (WTDS) | Days 1 and 28
PSG Total Sleep Time (TST) | Days 1 and 28
PSG Sleep Efficiency (SE) | Days 1 and 28
PSG Percent of Stages 1, 2, 3, 4 and REM sleep | Days 1 and 28
PSG Percent Slow Wave Sleep (SWS, Stages 3&4 combined) | Days 1 and 28
Subjective SL | Days 1 and 28
Subjective NA | Days 1 and 28
Subjective WASO | Days 1 and 28
Subjective TST | Days 1 and 28
Subjective ASR | Days 1 and 28
Subjective ASQ | Days 1 and 28
Karolinska Sleep Diary (KSD)-Sleep Quality Index | Days 1 and 28
KSD individual scores | Days 1 and 28
Vital signs | Days 1 and 28
Adverse events | Through Day 32

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Pfizer Investigational Site, Glendale, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Overland Park, Kansas

REFERENCES:
- [Derived] Furey SA, Hull SG, Leibowitz MT, Jayawardena S, Roth T. A randomized, double-blind, placebo-controlled, multicenter, 28-day, polysomnographic study of gabapentin in transient insomnia induced by sleep phase advance. J Clin Sleep Med. 2014 Oct 15;10(10):1101-9. doi: 10.5664/jcsm.4110. PMID 25317091
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A9451155&StudyName=A%2028-Day%20Polysomnographic%20Study%20of%20Gabapentin%20in%20Transient%20Insomnia%20Induced%20by%20a%20Sleep%20Phase%20Advance